CLINICAL TRIAL: NCT02580734
Title: Melatonin to Treat Burning Mouth Syndrome (BMS): A Randomized, Cross-over, Placebo-controlled, Triple-blind Clinical Trial
Brief Title: Efficacy of Melatonin in Burning Mouth Syndrome (BMS)
Acronym: BMS2013
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, ANDREA SARDELLA, Associate Professor of Oral Diseases, University of Milan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BMS2013
Record Dates: First submitted 2013-12-20; First posted 2015-10-20 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Burning Mouth Syndrome
Keywords: burning mouth syndrome; treatment; oral chronic pain
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): tablet without melatonin
  Interventions: Dietary Supplement: melatonin
- melatonin (Experimental): tablet with melatonin
  Interventions: Dietary Supplement: melatonin

INTERVENTIONS:
Dietary Supplement: melatonin — Cross-over randomized clinical trials

SUMMARY:
The purpose of this study is to determine whether melatonin is effective in the treatment of burning mouth syndrome (BMS).

DETAILED DESCRIPTION:
This is a crossover trial involving a total of 20 patients with Burning Mouth Syndrome, considered a chronic neuropathic pain. In two consecutive treatment periods, both 8 week long, each patient receives externally indistinguishable capsules (placebo or melatonin). A 4 weeks wash-out period is applied, between these two periods.

The capsules contain either placebo or 3 mg-melatonin (4 time/day for a total of 12 mg/day of melatonin). The primary endpoint is the change in pain intensity at the end of each treatment period, measured using VAS, verbal intensity score and NRS, as well as number of oral sites affected by the burning sensation. Furthermore, data from quality of life, anxiety and sleep questionnaires are collected (sf-36, HAM-A, ESS, MOS).

Adverse effects are carefully recorded as well as blood samples, in order to measure serum melatonin levels during the trial.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 yrs suffering from burning mouth syndrome

Exclusion Criteria:

* epilepsy
* pregnancy
* concomitant treatment with melatonin
* concomitant anticoagulants
* night time working persons

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Reduction/resolution of symptoms in BMS | within the first 60 days

SECONDARY OUTCOMES:
improvement in quality of life | within the first 60 days